CLINICAL TRIAL: NCT03123406
Title: A Multi-center Study Evaluating Efficacy and Safety of Cinacalcet Hydrochloride(HCL) in Calcium, Phosphorus and Intact Parathyroid Hormone(iPTH) Serum Levels in Chinese Chronic Kidney Disease(CKD) Hemodialysis(HD) Patients With Mild, Moderate and Severe Secondary Hyperparathyroidism(SHPT)
Brief Title: Efficacy and Safety of Cinacalcet in Ca, P and iPTH Levels in Patients With Mild, Moderate and Severe SHPT
Acronym: ACTIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyowa Kirin China Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKCN201601
Record Dates: First submitted 2017-03-29; First posted 2017-04-21 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hyperparathyroidism; Secondary, Renal
Keywords: cinacalcet; secondary hyperparathyroidism; calcimimetics; CKD-MBD
MeSH Terms: conditions — Hyperparathyroidism; Neoplasm Metastasis; Hyperparathyroidism, Secondary; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Cinacalcet

STUDY DESIGN:
Intervention Model Description: CKD Hemodialysis Patients with SHPT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Severe SHPT (Experimental): Administer Cinacalcet HCL to subjects whose iPTH>900 pg/ml from 1st to 32nd week.
  Interventions: Drug: Cinacalcet HCl
- Moderate SHPT (Experimental): Administer Cinacalcet HCL to subjects whose 600≤iPTH<900 pg/ml from 1st to 32nd week.
  Interventions: Drug: Cinacalcet HCl
- Mild SHPT (Experimental): Administer Cinacalcet HCL to subjects whose 300≤iPTH<600 pg/ml from 1st to 32nd week.
  Interventions: Drug: Cinacalcet HCl

INTERVENTIONS:
Drug: Cinacalcet HCl — Administer Cinacalcet HCL to all subjects from 1st to 32nd week. Subjects choose to buy and take Cinacalcet HCL in real-world period from 33rd to 52nd week.
  Other Names: Regpara

SUMMARY:
1. To evaluate achievement ratio of iPTH,Calcium and phosphorus after taking Cinacalcet HCL in hemodialysis subjects with mild, moderate and severe SHPT;
2. To explore the impact of Cinacalcet HCL using on the combined use of drugs;
3. To explore the difference of patients who continued or discontinued Cinacalcet HCL in real-world period from 33rd to 52nd week.

ELIGIBILITY:
Inclusion Criteria:

- Parents/guardians must sign informed consent;

Must be males or females whose age are 18 to 75 years old;

Clinical diagnosis of chronic kidney disease on maintenance hemodialysis with secondary hyperparathyroidism;

iPTH must be equal or higher than 300Pg/ml;

Must not have received Calcimimetics(for example, Cinacalcet) within 6 months prior to enrollment;

Must have been on maintenance hemodialysis 3 times weekly (TIW) for at least 3 months(12 weeks) prior to enrollment and must be expected to remain on hemodialysis for the duration of the study;

Over 2-year life expectancy.

Exclusion Criteria:

- Hypocalcemia [Corrected serum calcium level less than 2.1mmol/L(8.4mg/dL);

History of gastrointestinal bleeding or peptic ulcer disease and possibility of deterioration or recurrence;

Severe heart disease;

Epilepsy risk or history of epilepsy;

Hypersensitivity to Cinacalcet;

Drug abuse/addiction;

Plan to receive renal transplantation within 52 weeks;

Pregnant or lactating women;

Pregnancy plan within 1 years, or no guarantee on taking effective contraceptive measures within 1 year after enrollment;

Participated in other clinical trials within 4 weeks prior to enrollment;

Received parathyroidectomy within 24 weeks prior to enrollment;

Investigator judgment that patients are not suitable to enroll.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Compared with baseline data, the proportion of subjects reaching iPTH target at 20th week | 20 weeks
  blood test
Compared with baseline data, the proportion of subjects reaching iPTH target at 32nd week | 32 weeks
  blood test

SECONDARY OUTCOMES:
Compared with baseline data, the proportion of patients reaching Ca & P target simultaneously at 32nd week | 32 weeks
  blood test
Compared with baseline data, the proportion of patients with ≥ 30% reduction in iPTH level at 20th week | 20 weeks
  blood test
Compared with baseline data, the proportion of patients with ≥ 30% reduction in iPTH level at 32nd week | 32 weeks
  blood test
The proportion of patients once reaching iPTH target during 1st~32nd week | 32 weeks
  blood test
The proportion of patients once reaching iPTH target during 33rd~52nd week | 52 weeks
  blood test
Compared with baseline data, the change of Ca × P at 20th week | 20 weeks
  blood test
Compared with baseline data, the change of Ca × P at 32nd week | 32 weeks
  blood test
Compared with baseline data, the change of alkaline phosphatase (ALP) at 20th week | 20 weeks
  blood test
Compared with baseline data, the change of alkaline phosphatase (ALP) at 32nd week | 32 weeks
  blood test
Compared with baseline data, the change of fibroblast growth factor 23(FGF23) at 20th week | 20 weeks
  blood test
Compared with baseline data, the change of fibroblast growth factor 23(FGF23) at 32nd week | 32 weeks
  blood test
Compared with baseline data, the adjustment (type or amount) of calcium agents at 20th week | 20 weeks
  medication evaluation
Compared with baseline data, the adjustment (type or amount) of calcium agents at 32nd week | 32 weeks
  medication evaluation
Compared with baseline data, the adjustment (type or amount) of phosphate binders at 20th week | 20 weeks
  medication evaluation
Compared with baseline data, the adjustment (type or amount) of phosphate binders at 32nd week | 32 weeks
  medication evaluation
Compared with baseline data, the adjustment (type or amount) of vitamin D and its analogues at 20th week | 20 weeks
  medication evaluation
Compared with baseline data, the adjustment (type or amount) of vitamin D and its analogues at 32nd week | 32 weeks
  medication evaluation
Compared with baseline data, the adjustment (type or amount) of diphosphonic acid salts at 20th week | 20 weeks
  medication evaluation
Compared with baseline data, the adjustment (type or amount) of diphosphonic acid salts at 32nd week | 32 weeks
  medication evaluation
Compared with the data at 32nd week, the proportional change of patients reaching iPTH target at 52nd week who continue Cinacalcet treatment during 20-week real world period | 52 weeks
  blood test
Compared with the data at 32nd week, the proportional change of patients reaching iPTH target at 52nd week who discontinue Cinacalcet treatment after 20-week real world period | 52 weeks
  blood test
Compared with the data at 32nd week, the proportional change of patients reaching Ca target at 52nd week who continue Cinacalcet treatment after 20-week real world period | 52 weeks
  blood test
Compared with the data at 32nd week, the proportional change of patients reaching Ca target at 52nd week who discontinue Cinacalcet treatment after 20-week real world period | 52 weeks
  blood test
Compared with the data at 32nd week, the proportional change of patients reaching P target at 52nd week who continue Cinacalcet treatment after 20-week real world period | 52 weeks
  blood test
Compared with the data at 32nd week, the proportional change of patients reaching P target at 52nd week who discontinue Cinacalcet treatment after 20-week real world period | 52 weeks
  blood test
Compared with the data at 32nd week, the proportional change of patients reaching Ca × P target at 52nd week who continue Cinacalcet treatment after 20-week real world period | 52 weeks
  blood test
Compared with the data at 32nd week, the proportional change of patients reaching Ca × P target at 52nd week who discontinue Cinacalcet treatment after 20-week real world period | 52 weeks
  blood test
The dose change of calcium agents which were used by patients for chronic kidney disease-mineral and bone disorder(CKD-MBD) treatment during 20-week real world period | 20 weeks
  medication evaluation
The dose change of phosphate binders which were used by patients for chronic kidney disease-mineral and bone disorder(CKD-MBD) treatment during 20-week real world period | 20 weeks
  medication evaluation
The dose change of vitamin D and its analogues which were used by patients for chronic kidney disease-mineral and bone disorder(CKD-MBD) treatment during 20-week real world period | 20 weeks
  medication evaluation
The dose change of diphosphonic acid salts which were used by patients for chronic kidney disease-mineral and bone disorder(CKD-MBD) treatment during 20-week real world period | 20 weeks
  medication evaluation
The reasons of patients discontinuing Cinacalcet in 20-week real world | 20 weeks
  List presentation

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Study Chair — Jinling Hospital, China; Zhaohui Ni, Principal Investigator — RenJi Hospital; Zhangsuo Liu, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Jiazhuang Lou, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Guanqing Xiao, Principal Investigator — First People's Hospital of Foshan; Li Hao, Principal Investigator — The Second Hospital of Anhui Medial University; Ping Fu, Principal Investigator — West China Hopsital, Sichuan University; Yisheng Ling, Principal Investigator — Zhongshan Hospital Xiamen University; Xuemei Li, Principal Investigator — Peking Union Medical College Hospital; Shixiang Wang, Principal Investigator — Beijing Chao Yang Hospital; Aihua Zhang, Principal Investigator — Peking University Third Hospital; Xiaonong Chen, Principal Investigator — Ruijin Hospital; Jing Chen, Principal Investigator — Huashan Hospital; Li Zuo, Principal Investigator — Peking University People's Hospital; Aili Jiang, Principal Investigator — Tianjin Medical University Second Hospital; Guohua Ding, Principal Investigator — Hubei General Hospital; Jianying Niu, Principal Investigator — Fudan University; Yonghui Mao, Principal Investigator — Beijing Hospital; Qiang He, Principal Investigator — Sichuan Provincial People's Hospital; Chaosheng Chen, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; Hong Liu, Principal Investigator — Second Xiangya Hospital of Central South University; Junwei Yang, Principal Investigator — Second Affiliated Hospital of Nanjing Medical University; Jianming Ye, Principal Investigator — The First People's Hospital of Kunshan
Locations (1):
- Nanjing Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided